CLINICAL TRIAL: NCT02430584
Title: Whole Blood Specimen Collection From Pregnant Subjects
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progenity, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-101-SAMPLES
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Down Syndrome; Edwards Syndrome; Patau Syndrome; Klinefelter Syndrome; Turner Syndrome; DiGeorge Syndrome; Perinatal Infections
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Klinefelter Syndrome; Turner Syndrome; DiGeorge Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Study will collect up to 50 mL of whole blood at one or more monthly clinic visits (≥25 days apart) from pregnant women carrying a single fetus of 10 to 26 weeks of gestational age
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational - no intervention

SUMMARY:
To obtain whole blood specimens from pregnant subjects to be used for research and development and clinical validation studies of prenatal assays.

DETAILED DESCRIPTION:
This sample collection protocol allows for the identification, recruitment, and participation in women who are pregnant and are known to:

1. be at an increased risk for fetal genetic abnormalities
2. be at increased risk for congenital fetal infection by virtue of being positive by initial screening tests, or are known to have an active infection during this pregnancy.
3. possess irregular blood group antigens (the subject or the father of the baby) and are therefore at increased risk for fetal sensitization during this pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing to provide consent to have up to 50 mL of whole blood collected at one or more monthly (≥25 days) clinic visits
* Subject is pregnant carrying a singleton fetus of 10 to 26 weeks gestational age inclusive
* Subject is 18 years of age or older
* Subject is at an increased risk for one or more of the following:

  * fetal gene and chromosome abnormalities
  * congenital fetal infection
  * known to possess irregular blood group antigens (subject or father of the baby)
  * known to have some other condition amenable to noninvasive prenatal testing

Exclusion Criteria:

* Pregnancy is non-viable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: GENDER: Female ETHNICITY: All ethnicities RACE: All races AGE: Subjects 18 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Whole blood collection | One or more monthly clinic visits (≥25 days apart) over 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Obstetrical Consultants, Chattanooga, Tennessee, United States